CLINICAL TRIAL: NCT05480878
Title: Clinical Study Evaluating the Efficacy of Nitazoxanide and Escitalopram as Adjuvant Therapies in Patients With Rheumatoid Arthritis
Brief Title: Role of Nitazoxanide and Escitalopram in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Abeer Abdelmhsen Elsayed Elmotwally, Assistant lecturer at clinical pharmacy department ,faculty of pharmacy, Tanta university, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rheumatoid Arthritis
Record Dates: First submitted 2022-07-23; First posted 2022-07-29 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Nitazoxanide; Escitalopram; STAT3/ JAK2 signaling pathway; TLR-4 /IL -1β signaling pathway
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — nitazoxanide; Tablets; Escitalopram

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): Participants in this arm will receive Placebo with the current DMARDs treatments for rheumatoid arthritis for 12 weeks.
  .
  Interventions: Drug: Placebo
- Nitazoxanide (Experimental): Participants in this arm will receive Nitazoxanide 1 gm/day + DMARDs for 12 weeks.
  Interventions: Drug: Nitazoxanide 500Mg Oral Tablet
- Escitalopram (Experimental): Participants in this arm will receive Escitalopram 10 mg/day + DMARDs for 12 weeks.
  Interventions: Drug: Escitalopram 10mg

INTERVENTIONS:
Drug: Placebo — Placebo will be administered to the control group for 12 weeks as an add-on treatment to the current DMARDs treatments for rheumatoid arthritis.
  Arms: Control
Drug: Nitazoxanide 500Mg Oral Tablet — All subjects will receive Nitazoxanide 500gm twice daily for 12 weeks as an add-on treatment to the current DMARDs treatments for rheumatoid arthritis.
  Arms: Nitazoxanide
Drug: Escitalopram 10mg — All subjects will receive Escitalopram 10 mg/day for 12 weeks as an add-on treatment to the current DMARDs treatments for rheumatoid arthritis.
  Arms: Escitalopram

SUMMARY:
This study aims at evaluating the therapeutic effects of both Nitazoxanide and Escitalopram as adjuvant therapies in patients with Rheumatoid Arthritis and to evaluate their impact on STAT3/ JAK2, TLR /IL -1β signaling pathways.

DETAILED DESCRIPTION:
This study is a randomized, controlled prospective study to evaluate the potential therapeutic effects of the broad -spectrum antimicrobial (Nitazoxanide) and selective serotonin reuptake inhibitor (Escitalopram) on synovial inflammation and angiogenesis when administered as add-on treatments to the current DMARDs treatments for rheumatoid arthritis patients.

A total of 90 RA patients recruited from Outpatient Clinic of Physical Medicine, Rheumatology and Rehabilitation at Mansoura University hospitals, Mansoura, Egypt will be included in the study. They will be diagnosed with RA according to the American College of Rheumatology/European League Against Rheumatism criteria 2010 (the ACR/EULAR 2010 criteria).

RA Patients who will meet the inclusion criteria will be enrolled in the study.

They will be classified into three groups:

Group 1: 30 RA patients who will receive the traditional therapy of rheumatoid arthritis for 12 weeks and serve as the control group.

Group 2: 30 RA patients who will receive traditional therapy plus Nitazoxanide 1 gm/day for 12 weeks.

Group 3: 30 RA patients who will receive traditional therapy plus Escitalopram 10 mg/day for 12 weeks.

Clinical Examinations and laboratory parameters will be performed and measured at the beginning of the study and 3 months after randomization to evaluate the efficacy of Nitazoxanide and Escitalopram in the treatment of rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis according to the ACR/EULAR 2010 criteria.
* Receiving conventional disease modified anti rheumatic drugs (DMARDS).
* Having active disease (the 28-joint disease activity score [DAS28] according to the CRP formula > 2.6).
* Age between 18 and 75 years.
* Conscious and cooperative.
* Male or female.
* Sign an informed consent for the clinical study

Exclusion Criteria:

1. Pregnant or planning to be pregnant and breast-feeding women.
2. Chronic disease.
3. Other autoimmune diseases, such as systemic lupus erythematosus, Sjogren's syndrome and mixed connective tissue disease.
4. Patients treated with biological TNF-α, IL6 or IL-1β antagonists.
5. Infectious or inflammatory diseases, endocrine disorders, any past or current psychiatric or neurological diseases.
6. Clinically significant hepatic and renal dysfunction or impairment.
7. Alcohol abuse
8. Receiving therapy that interact with Nitazoxanide and Escitalopram.
9. Hypersensitivity to Nitazoxanide and Escitalopram.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in Clinical Disease Activity Index (CDAI) Score | Baseline, 12 weeks
  To evaluate the effect of the use of Nitazoxanide and Escitalopram as an add-on therapy in patients with rheumatoid arthritis by evaluating the change from baseline in the clinical findings as measured by Clinical Disease Activity Index (CDAI) scores. A lower CDAI score from Baseline would mean improvement in disease activity and an increase in CDAI score from Baseline would mean an increase in disease activity or a worsening in disease activity. Scores: 0.0-2.8 = Range for Remission; 2.9-10.0 = Range for Low disease activity; 10.1-22.0 Range for Moderate disease activity; 22.1-76 Range for High disease activity. Total range is from 0-100, with the high scores representing high disease activity.
Changes in Erythrocyte Sedimentation Rates (ESR) | Baseline, 12 weeks
  Erythrocyte Sedimentation Rates (ESR) values will be made at baseline and after 12 weeks to determine the number of patients whose test result improved or worsened. ESR (normal range 0-28 mm/hr). If the value is increased, the disease activity worsened. If the value is reduced the disease activity is improved.
Changes in C- reactive Protein (CRP) | Baseline,12 weeks
  C- reactive Protein (CRP) values will be made at baseline and after 12 weeks to determine the number of patients whose test result improved or worsened. CRP value (normal range <1.0 mg/dl). If the value is increased, the disease activity worsened. If the value is reduced the disease activity is improved.
Changes in Rheumatoid factor (RF) values | Baseline,12 weeks
  Rheumatoid factor (RF) values will be made at baseline and after 12 weeks to determine the number of patients whose test result improved or worsened. If the value is increased, the disease activity worsened. If the value is reduced the disease activity is improved.
Changes in Anti-cyclic citrullinated peptide (Anti-CCP) values | Baseline,12 weeks
  Anti-cyclic citrullinated peptide (Anti-CCP) values will be made at baseline and after 12 weeks to determine the number of patients whose test result improved or worsened. If the value is increased, the disease activity worsened. If the value is reduced the disease activity is improved.

SECONDARY OUTCOMES:
Determination of Signal transducer and activator of transcription 3 (STAT3) levels | Baseline,12 weeks
  Serum STAT3 levels will be measured by means of the human enzyme-linked immunosorbent assay (ELISA) technique according to the manufacturers protocol
Determination of Toll-like receptor4 (TLR-4) levels | Baseline,12 weeks
  Serum TLR4 levels will be measured by means of the human enzyme-linked immunosorbent assay (ELISA) technique according to the manufacturers protocol.
Determination of interleukin-1β (IL-1β) levels | Baseline, 12 weeks
  Serum IL-1β levels will be measured by means of the human enzyme-linked immunosorbent assay (ELISA) technique according to the manufacturers protocol.
Determination of Malondialdehyde (MDA) levels | Baseline, 12 weeks
  Serum MDA levels will be measured by means of the human enzyme-linked immunosorbent assay (ELISA) technique according to the manufacturers protocol

OTHER OUTCOMES:
Numbers of participants with treatment-related adverse events | Baseline, 12 weeks
  The adverse events in each group will be observed and documented during the whole procedure to show the safety of the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smolen JS, Aletaha D, Barton A, Burmester GR, Emery P, Firestein GS, Kavanaugh A, McInnes IB, Solomon DH, Strand V, Yamamoto K. Rheumatoid arthritis. Nat Rev Dis Primers. 2018 Feb 8;4:18001. doi: 10.1038/nrdp.2018.1. PMID 29417936
- [Background] Li Y, de Haar C, Peppelenbosch MP, van der Woude CJ. New insights into the role of STAT3 in IBD. Inflamm Bowel Dis. 2012 Jun;18(6):1177-83. doi: 10.1002/ibd.21884. Epub 2011 Oct 12. PMID 21994179
- [Background] Wu X, Shou Q, Chen C, Cai H, Zhang J, Tang S, Cai B, Tang D, Cao G. An herbal formula attenuates collagen-induced arthritis via inhibition of JAK2-STAT3 signaling and regulation of Th17 cells in mice. Oncotarget. 2017 Jul 4;8(27):44242-44254. doi: 10.18632/oncotarget.17797. PMID 28562338
- [Background] Aboudounya MM, Heads RJ. COVID-19 and Toll-Like Receptor 4 (TLR4): SARS-CoV-2 May Bind and Activate TLR4 to Increase ACE2 Expression, Facilitating Entry and Causing Hyperinflammation. Mediators Inflamm. 2021 Jan 14;2021:8874339. doi: 10.1155/2021/8874339. eCollection 2021. PMID 33505220
- [Background] Li CH, Lu ZR, Zhao ZD, Wang XY, Leng HJ, Niu Y, Wang MP. Nitazoxanide, an Antiprotozoal Drug, Reduces Bone Loss in Ovariectomized Mice by Inhibition of RANKL-Induced Osteoclastogenesis. Front Pharmacol. 2021 Dec 9;12:781640. doi: 10.3389/fphar.2021.781640. eCollection 2021. PMID 34955850
- [Background] Lu Z, Li X, Li K, Wang C, Du T, Huang W, Ji M, Li C, Xu F, Xu P, Niu Y. Structure-Activity Study of Nitazoxanide Derivatives as Novel STAT3 Pathway Inhibitors. ACS Med Chem Lett. 2021 Apr 1;12(5):696-703. doi: 10.1021/acsmedchemlett.0c00544. eCollection 2021 May 13. PMID 34055214
- [Background] Gong F, Shen T, Zhang J, Wang X, Fan G, Che X, Xu Z, Jia K, Huang Y, Li X, Lu H. Nitazoxanide induced myocardial injury in zebrafish embryos by activating oxidative stress response. J Cell Mol Med. 2021 Oct;25(20):9740-9752. doi: 10.1111/jcmm.16922. Epub 2021 Sep 17. PMID 34533278
- [Background] Sacre S, Medghalchi M, Gregory B, Brennan F, Williams R. Fluoxetine and citalopram exhibit potent antiinflammatory activity in human and murine models of rheumatoid arthritis and inhibit toll-like receptors. Arthritis Rheum. 2010 Mar;62(3):683-93. doi: 10.1002/art.27304. PMID 20131240
- [Background] Gupta S, Upadhayay D, Sharma U, Jagannathan NR, Gupta YK. Citalopram attenuated neurobehavioral, biochemical, and metabolic alterations in transient middle cerebral artery occlusion model of stroke in male Wistar rats. J Neurosci Res. 2018 Jul;96(7):1277-1293. doi: 10.1002/jnr.24226. Epub 2018 Apr 15. PMID 29656429
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Nishimoto N, Takagi N. Assessment of the validity of the 28-joint disease activity score using erythrocyte sedimentation rate (DAS28-ESR) as a disease activity index of rheumatoid arthritis in the efficacy evaluation of 24-week treatment with tocilizumab: subanalysis of the SATORI study. Mod Rheumatol. 2010 Dec;20(6):539-47. doi: 10.1007/s10165-010-0328-0. Epub 2010 Jul 10. PMID 20617358